CLINICAL TRIAL: NCT00323947
Title: Double Blind, Placebo Controlled, Crossover Study of Extended Release Methylphenidate for Treatment of ADHD in Children With Epilepsy
Brief Title: Methylphenidate for Treating Attention Deficit Hyperactivity Disorder in Children With Both ADHD and Epilepsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K23MH066835 (NIH); K23MH066835 (NIH); DDTR BK-TKND
Record Dates: First submitted 2006-05-08; First posted 2006-05-10 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Epilepsy
Keywords: ADHD; Seizures; Methylphenidate; Stimulant
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Epilepsy; Seizures | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Participants will take OROS-MPH then switch to placebo
  Interventions: Drug: Extended Release Methylphenidate (OROS-Methylphenidate)
- 2 (Placebo Comparator): Participants will take placebo then switch to OROS-MPH
  Interventions: Drug: Extended Release Methylphenidate (OROS-Methylphenidate)

INTERVENTIONS:
Drug: Extended Release Methylphenidate (OROS-Methylphenidate) — Participants will first take either immediate release MPH or placebo "A" for 1 day. On Day 2 of treatment, participants assigned to receive XR-MPH will begin taking it, and participants assigned to receive placebo will switch to placebo "B." This treatment phase will continue for 6 days to 4 weeks, depending on weight, and will then be followed by a 1-week medication washout period. Target dose depends on the weight of the participant. Possible dose forms include 18, 36, 54 mg OROS-MPH.
  Other Names: Concerta

SUMMARY:
This study will evaluate the safety and effectiveness of extended release methylphenidate (XR-MPH) in treating attention deficit hyperactivity disorder (ADHD) in children with both ADHD and epilepsy.

DETAILED DESCRIPTION:
Epilepsy is a brain disorder in which clusters of nerve cells in the brain periodically send abnormal signals. The normal pattern of nerve cell activity, therefore, becomes disrupted, which can result in seizures. Some symptoms of epileptic seizures include the following: strange sensations, emotions, or behavior; convulsions; muscle spasms; and loss of consciousness. Children with epilepsy are at risk for other specific disorders, such as ADHD, one of the most common mental disorders in children. ADHD is characterized by impulsiveness, hyperactivity, and inattention. Approximately one third of children with epilepsy also have ADHD. Stimulant medication is a common treatment method for ADHD. The effect of stimulant treatment on epilepsy and seizure frequency, however, is unknown. This study will evaluate the safety and effectiveness of XR-MPH, a stimulant medication, in treating ADHD in children with both ADHD and epilepsy.

People interested in participating in this double-blind study will first attend two visits for interviews and evaluations to determine eligibility for participation. Upon study entry, participants will be randomly assigned to initially receive either XR-MPH or placebo. Medication dosages and duration in the study will depend on participants' weights. Participants will first take either immediate release MPH or placebo "A" for 1 day. Any participants who experience an adverse event will be removed from the study. On Day 2 of treatment, participants assigned to receive XR-MPH will begin taking it, and participants assigned to receive placebo will switch to placebo "B." This treatment phase will continue for 6 days to 4 weeks, depending on weight, and will then be followed by a 1-week medication washout period. Following the washout, participants will switch to the other treatment group for the remainder of the study and will receive either XR-MPH or placebo in the same manner. Participants will attend weekly study visits, at which they will receive medication and undergo assessments of ADHD symptoms and medication side effects. Blood will be drawn to assess medication levels at the first study visit and following both rounds of treatment. Participants who have trouble with transportation to and from the study site may complete some study visits via telephone. Upon study completion, all participants will be offered clinical treatment with the study physician. Follow-up visits will be held every 2 to 6 months for patients who choose to continue receiving care from the study physician.

ELIGIBILITY:
Inclusion Criteria:

* Speaks English
* Intelligence Quotient (IQ) of greater than 35 and scores greater than 35 on the Scales of Independent Behavior - Revised (SIB-R) Broad Independence Scale (both IQ and adaptive functioning at the Moderate Mental Retardation level or higher)
* Diagnosis of epilepsy by International League Against Epilepsy (ILEA) criteria 26 (repeated, afebrile, unprovoked seizures with a seizure within the past 5 years)
* Diagnostic and Statistical Manual (DSM)-IV diagnosis of ADHD
* Scores at least 4 on the CGI severity scale for ADHD
* Scores greater than 90% on the ADHD Rating Scale (ADHD RS), Parent Version; investigator scored for age and sex on either the inattentive, hyperactive-impulsive, or total score at first visit
* Has not taken stimulants or alpha-adrenergic medications for more than 2 weeks prior to study entry
* If taking antidepressants, neuroleptics, or lithium, doses have been stable for more than 4 weeks
* Currently on an antiepileptic drug (AED) regimen with stable doses for more than 4 weeks prior to study entry
* Seizure-free for more than 1 month prior to study entry
* Prescribing clinician for epilepsy anticipates the need for a stable AED regimen for the duration of the study
* Guardian gives permission for study personnel to communicate with prescribing epilepsy clinician
* Teacher agrees to fill out ADHD RS at baseline and at the end of each arm of the study

Exclusion Criteria:

* Has had a seizure within the month preceding study entry
* Change in AED regimen or dose within 4 weeks of study entry
* History of moderate or severe adverse event related to MPH
* History of any psychotic disorder
* Current acute major depression or bipolar mania
* Current psychiatric disorder requiring pharmacotherapy (other than ADHD)
* Unstable significant medical condition other than epilepsy
* Any known conditions that may make treatment with MPH medically inadvisable
* Not currently working with a physician for epilepsy treatment
* Previously participated in a trial that provided adequate treatment with XR-MPH
* Weighs less than 9 kg
* Pregnant
* Unwilling to use an effective form of contraception
* Child has taken a stimulant (MPH, an amphetamine preparation, or pemoline), alpha-adrenergic (clonidine or guanfacine), or other ADHD medication within 2 weeks of the screening telephone interview. Children will not be withdrawn from psychotropic medications in order to be enrolled in the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2003-05; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Seizure occurence | Measured between Weeks 1 and 4
Clinical administered scores on the ADHD Rating Scale IV Parent Version | Measured between Weeks 1 and 4

SECONDARY OUTCOMES:
CGI-ADHD-Severity | Measured between Weeks 1 and 4
ADHD Rating Scale IV Teacher Version | Measured between Weeks 1 and 4
Scores on the Barkley Side Effects Checklist-Modified | Measured between Weeks 1 and 4
Clinical Global Impressions (CGI)-ADHD-Improvement | Measured between Weeks 1 and 4

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M. Gonzalez-Heydrich, MD, Principal Investigator — Children's Hospital Boston, Harvard Medical School
Locations (1):
- Childrens Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Eaton C, Yong K, Walter V, Mbizvo GK, Rhodes S, Chin RF. Stimulant and non-stimulant drug therapy for people with attention deficit hyperactivity disorder and epilepsy. Cochrane Database Syst Rev. 2022 Jul 13;7(7):CD013136. doi: 10.1002/14651858.CD013136.pub2. PMID 35844168